CLINICAL TRIAL: NCT02859558
Title: Effect of Antiretroviral Treatment Initiated During Acute HIV-1 Infection on Measures of HIV-1 Persistence and on HIV-1-Specific Immune Responses
Brief Title: Early ART to Limit Infection and Establishment of Reservoir
Acronym: EARLIER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5354; 2UM1AI068636 (NIH)
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Results first posted 2022-01-03 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — elvitegravir; bictegravir, emtricitabine, tenofovir alafenamide, drug combination; Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Fiebig I/II (Experimental): Participants enrolled during Fiebig stages I or II (non-reactive HIV-1 antibody).
  Interventions: Drug: elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide or bictegravir/emtricitabine/tenofovir alafenamide or other medically-appropriate FDA-approved antiretroviral therapy
- Arm 2: Fiebig III/IV (Experimental): Participants enrolled during Fiebig stages III or IV (reactive HIV-1 antibody and negative or indeterminate results on the Western blot or Geenius HIV-1/HIV-2).
  Interventions: Drug: elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide or bictegravir/emtricitabine/tenofovir alafenamide or other medically-appropriate FDA-approved antiretroviral therapy
- Arm 3: Fiebig V (Experimental): Participants enrolled during Fiebig stage V (reactive HIV-1 antibody and positive Western blot or Geenius HIV-1/HIV-2 without p31 band).
  Interventions: Drug: elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide or bictegravir/emtricitabine/tenofovir alafenamide or other medically-appropriate FDA-approved antiretroviral therapy

INTERVENTIONS:
Drug: elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide or bictegravir/emtricitabine/tenofovir alafenamide or other medically-appropriate FDA-approved antiretroviral therapy — Participants received one tablet of elvitegravir 150mg/cobicistat 150mg/emtricitabine 200mg/tenofovir alafenamide 10mg by mouth daily with food or one tablet of bictegravir 50mg/emtricitabine 200mg/tenofovir alafenamide 25mg by mouth daily with or without food. Other non-study-provided ARV regimens were allowed for participants who were pregnant, breastfeeding, or unable/unwilling to take EVG/COBI/FTC/TAF or BIC/FTC/TAF, or for participants whose local health care/primary care provider preferred starting a different initial ARV regimen.
  Other Names: Single-tablet regimen EVG/COBI/FTC/TAF or Genvoya; Single-tablet regimen BIC/FTC/TAF or Biktarvy

SUMMARY:
The study was done to:

* Start antiretroviral therapy (ART) early in those recently or acutely infected with HIV-1
* See how starting ART as soon as the infection is found affects the amount of HIV-1 in blood and how well the body fights the HIV-1 infection
* Look at the amount of HIV-1 DNA (genetic material for HIV-1) seen in CD4+ T-cells (infection-fighting cells in blood) after 48 weeks of ART
* See how early treatment for HIV affects the numbers of HIV-1 infection fighting cells (CD4+ and CD8+ T-cells) in blood

DETAILED DESCRIPTION:
This was a Phase II, prospective, open-label two-step study to measure the effects of early ART on the establishment of HIV-1 reservoir and HIV-1-specific immunity. Participants were enrolled if they fulfilled the inclusion criteria for acute HIV-1 infection (AHI) diagnosis within 7 days prior to entry and had an enrollment visit with the immediate initiation of ART. Plasma and serum samples for Fiebig staging were collected at the time of ART initiation.

Participants were followed for up to 216 weeks (72 weeks on Step 1 and 144 weeks on Step 2). Evaluations at weeks 2 and 8 on Step 1 were performed via telephone.

The Fiebig stage-classification system was used to characterize the progression from HIV-1 exposure to HIV-1 seroconversion at the time of ART initiation. In this study, the five Fiebig stages of interest were simplified into three study groups as described below (based on HIV-1 antibody diagnostic profile at time of ART initiation).

The primary analysis was based on Step 1. Step 2 was added to the study for long term follow-up. The rationale for the extended follow-up period was to expand the number of available participants for future therapeutic and cure studies without the burden of frequent visits and the cost of study-provided laboratory testing.

Group 1: Fiebig I/II (non-reactive HIV-1 antibody)

Group 2: Fiebig III/IV (reactive HIV-1 antibody and negative or indeterminate results on the Western Blot (WB) or Geenius HIV-1/HIV-2)

Group 3: Fiebig V (reactive HIV-1 antibody and positive WB or Geenius HIV-1/HIV-2 without p31 band)

Although participants in Fiebig VI (positive WB or Geenius HIV-1/HIV-2 with p31 band) were not specifically targeted for enrollment in this study, it was possible that a small number of participants would be determined to be in Fiebig VI (positive Western blot or Geenius HIV-1/HIV-2 with p31 band) based on analysis of the entry samples. Participants who were determined to be in Fiebig VI were followed on the study for no more than 24 weeks on Step 1, allowing ample time for them to pursue alternative sources for ART. Enrolled participants without HIV or in Fiebig VI were replaced.

The study-provided regimen was single tablet regimen elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (EVG/COBI/FTC/TAF) or bictegravir/emtricitabine/tenofovir alafenamide (BIC/FTC/TAF). Other non-study-provided antiretroviral (ARV) regimens were also allowed for participants who were pregnant, breastfeeding, or unable/unwilling to take EVG/COBI/FTC/TAF or BIC/FTC/TAF, or for participants whose local health care/primary care provider preferred starting a different initial ARV regimen.

ELIGIBILITY:
Inclusion Criteria:

Appropriate documentation from medical records of diagnosis of acute HIV-1 infection (AHI) within 7 days prior to enrollment, that includes one of the following:

1. A detectable HIV-1 RNA within 28 days prior to study entry AND a non-reactive HIV-1 antibody within 7 days prior to entry OR
2. A detectable HIV-1 RNA or a reactive HIV-1 antibody within 28 days prior to study entry AND a negative/indeterminate WB or negative/indeterminate Geenius HIV-1/HIV-2 Supplemental Assay within 7 days prior to entry OR
3. A documented non-reactive HIV-1 antibody or negative HIV-1 RNA within 90 days prior to study entry AND a documented reactive HIV-1 antibody or positive WB that is negative for p31 band or a positive Geenius HIV-1/HIV-2 Supplemental Assay that is negative for p31 band within 7 days prior to entry OR
4. ARCHITECT or GSCOMBO S/CO ≥10 within 7 days prior to entry AND a non-reactive HIV-1 antibody within 7 days prior to entry OR
5. ARCHITECT or GSCOMBO S/CO ≥1 within 7 days prior to entry AND a non-reactive HIV-1 antibody within 7 days prior to entry AND a known prior S/CO <0.5 within 90 days prior to entry OR
6. ARCHITECT or GSCOMBO S/CO >0.5 but <10 within 7 days prior to entry AND a non-reactive HIV-1 antibody within 7 days prior to entry AND detectable HIV-1 RNA within 7 days prior to entry

Note A: HIV-1 RNA result must be reported from an FDA-approved or CE-marked assay.

Note B: Since characterization of Fiebig stage using samples at the time of ART initiation was performed with results known within 12 weeks based on standardized, centralized testing, an estimated Fiebig group at enrollment based on inclusion criteria as shown in the table above will provide additional real-time monitoring for accruals into each study group.

* Ability and willingness of candidate to provide written informed consent.
* Ability and willingness to initiate ART at enrollment.
* Ability and willingness to participate in scheduled study visits for up to 72 weeks.
* Female candidates of reproductive potential who are not pregnant at the time of enrollment and who will receive the study-provided EVG/COBI/FTC/TAF and must agree not to participate in the conception process (ie, active attempt to become pregnant, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, the female candidate must agree to use at least one reliable form of contraceptive while receiving study-provided treatment.

Female candidates are considered to be of reproductive potential if any of the following conditions apply:

* Candidate has experienced menarche.
* Candidate has not undergone bilateral tubal ligation, bilateral oophorectomy, or hysterectomy.
* Candidate has not experienced menopause, defined as lack of menstruation within the preceding 12 months.

Acceptable contraceptive methods include:

* Condoms (male or female) with or without a spermicidal agent
* Diaphragm or cervical cap with spermicide
* Intrauterine device
* Hormonal contraceptive

Female candidates who are not of reproductive potential or whose male partner(s) has documented azoospermia are not required to use contraceptives. Any statement of self-reported sterility or that of her partner must be entered in the source documents.

NOTE: Acceptable documentation of lack of reproductive potential is oral or written documentation from the individual.

Female candidates who are prescribed a non-study-provided ARV regimen should discuss the safety of that regimen during conception and pregnancy with the prescribing physician. Such individuals should follow medical guidance regarding any potential need for contraception while using the non-study-provided ARV regimen.

Note: Pregnant and breastfeeding women may enroll in the study provided that they meet the eligibility requirements and have access to non-study-provided ARV regimens.

Exclusion Criteria:

* Positive HIV-1 antibody test ≥90 days prior to study entry.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Any acute, chronic, or recent and clinically significant medical condition that, in the opinion of the site investigator, would interfere with adherence to study requirements or jeopardize the safety or rights of the participant.
* Receipt of an investigational study agent within 28 days prior to enrollment
* Chronic or recurrent use of medications that modify host immune response, eg, oral or parenteral steroids, cancer chemotherapy.
* AHI diagnosis within 60 days after receiving any investigational ARV or HIV-1 vaccine or immune prophylaxis for HIV-1 infection.
* Use of ARVs for pre- or post-exposure prophylaxis within 60 days prior to the diagnosis of AHI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2025-04-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (23):
  - 31788 Alabama CRS, Birmingham, Alabama
  - Ucsd, Avrc Crs (701), San Diego, California
  - Harbor-UCLA Med. Ctr. CRS (603), Torrance, California
  - Whitman Walker Health CRS (31791), Washington D.C., District of Columbia
  - The Ponce de Leon Center CRS (5802), Atlanta, Georgia
  - Northwestern University CRS (2701), Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS (2702), Chicago, Illinois
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS (107), Boston, Massachusetts
  - Washington University CRS (2101), St Louis, Missouri
  - 31786 New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - 7804 Weill Cornell Chelsea CRS, New York, New York
  - Columbia Physicians and Surgeons CRS (30329), New York, New York
  - 3201 Chapel Hill CRS, Chapel Hill, North Carolina
  - Greensboro CRS (3203), Greensboro, North Carolina
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - The Ohio State Univ. AIDS CRS (2301), Columbus, Ohio
  - 6201 Penn Therapeutics CRS, Philadelphia, Pennsylvania
  - Pittsburgh CRS (1001), Pittsburgh, Pennsylvania
  - The Miriam Hosp. ACTG CRS (2951), Providence, Rhode Island
  - 31443 Trinity Health and Wellness Center CRS, Dallas, Texas
  - 31473 Houston AIDS Research Team (HART) CRS, Houston, Texas
  - University of Washington AIDS CRS (1401), Seattle, Washington
- Brazil (2):
  - Hospital Nossa Senhora da Conceicao CRS (12201), Porto Alegre, Rio Grande do Sul
  - Instituto de Pesquisa Clinica Evandro Chagas (12101), Rio de Janeiro
- Malawi CRS (12001), Lilongwe, Malawi
- Peru (2):
  - San Miguel CRS (11302), San Isidro, Lima region
  - Barranco CRS, Lima
- 31802 Thai Red Cross AIDS Research Center Treatment (TRC-ARC Treatment) CRS, Bangkok, Patumwan, Thailand
- Milton Park CRS (30313), Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the Advancing Clinical Therapeutics Globally (ACTG) by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the ACTG.
  * For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the ACTG "Data Request" form at: https://actgnetwork.org/submit-a-proposal/. Researchers of approved proposals will need to sign an ACTG Data Use Agreement before receiving the data.

REFERENCES:
- [Derived] Crowell TA, Ritz J, Coombs RW, Zheng L, Eron JJ, Mellors JW, Dragavon J, van Zyl GU, Lama JR, Ruxrungtham K, Grinsztejn B, Arduino RC, Fox L, Ananworanich J, Daar ES; AIDS Clinical Trials Group A5354/EARLIER (Early ART to Limit Infection and Establishment of Reservoir) Study Team. Novel Criteria for Diagnosing Acute and Early Human Immunodeficiency Virus Infection in a Multinational Study of Early Antiretroviral Therapy Initiation. Clin Infect Dis. 2021 Aug 2;73(3):e643-e651. doi: 10.1093/cid/ciaa1893. PMID 33382405
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 2.1, July 2017 — http://rsc.tech-res.com/clinical-research-sites/safety-reporting/daids-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from January 2017 to December 2019 at 30 sites in Brazil, Malawi, Peru, Thailand, United States, and Zimbabwe.
Pre-assignment Details: There was no randomization in this study. Participants who were determined to be in Fiebig VI were followed on the study for no more than 24 weeks on Step 1. Confirmed Fiebig VI and HIV negative participants were replaced.
Groups:
- Fiebig VI: Participants enrolled during Fiebig stage VI (reactive HIV-1 antibody and positive Western blot or Geenius HIV-1/HIV-2 without p31 band).
  elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide or bictegravir/emtricitabine/tenofovir alafenamide or other medically-appropriate FDA-approved antiretroviral therapy: Participants received one tablet of elvitegravir 150mg/cobicistat 150mg/emtricitabine 200mg/tenofovir alafenamide 10mg by mouth daily with food or one tablet of bictegravir 50mg/emtricitabine 200mg/tenofovir alafenamide 25mg by mouth daily with or without food. Other non-study-provided ARV regimens were allowed for participants who were pregnant, breastfeeding, or unable/unwilling to take EVG/COBI/FTC/TAF or BIC/FTC/TAF, or for participants whose local health care/primary care provider preferred starting a different initial ARV regimen.
- HIV-negative: Participants found to be HIV negative following the results of HIV-1 RNA testing at study entry. No study treatment.
Period: Step 1
Arm/Group | Arm 1: Fiebig I/II | Arm 2: Fiebig III/IV | Arm 3: Fiebig V | Fiebig VI | HIV-negative
Started | 49 | 79 | 60 | 4 | 3
Completed Week 48 | 41 | 68 | 50 | 0 | 0
Completed | 37 | 67 | 49 | 4 | 0
Not Completed | 12 | 12 | 11 | 0 | 3
Not completed — Not Eligible | 0 | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 1 | 3 | 3 | 0 | 0
Not completed — Did Not Return to Clinic | 2 | 3 | 4 | 0 | 0
Not completed — Moved | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal By Participant | 1 | 2 | 1 | 0 | 0
Not completed — Had to Interrupt antiretroviral (ARV) | 1 | 0 | 0 | 0 | 0
Not completed — Incarceration | 0 | 1 | 0 | 0 | 0
Not completed — Non-Adherence to Study Drug | 2 | 0 | 1 | 0 | 0
Not completed — Non-Adherence to Study Requirements | 3 | 1 | 0 | 0 | 0
Not completed — Virologic Failure | 2 | 1 | 1 | 0 | 0
Period: Step 2
Arm/Group | Arm 1: Fiebig I/II | Arm 2: Fiebig III/IV | Arm 3: Fiebig V | Fiebig VI | HIV-negative
Started (Some participants who completed Step 1 did not enroll to Step 2.) | 26 | 42 | 23 | 0 | 0
Completed | 22 | 37 | 19 | 0 | 0
Not Completed | 4 | 5 | 4 | 0 | 0
Not completed — Lost to Follow-up | 3 | 3 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0
Not completed — Unexpected Closure of Site | 0 | 1 | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Incarceration | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants with available baseline measurements.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Fiebig I/II | Arm 2: Fiebig III/IV | Arm 3: Fiebig V | Fiebig VI | HIV-negative | Total
Number analyzed (Participants) | 49 | 79 | 60 | 4 | 3 | 195
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [22 to 35] | 30 [24 to 40] | 26 [23 to 38] | 36 [22 to 48] | 25 [19 to 39] | 27 [23 to 39]
Age, Customized [Count of Participants; unit: Participants]
  18-29 years | 31 | 39 | 36 | 2 | 2 | 110
  30-39 years | 12 | 18 | 12 | 0 | 1 | 43
  40-49 years | 4 | 12 | 6 | 2 | 0 | 24
  50+ years | 2 | 10 | 6 | 0 | 0 | 18
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Cisgender | 47 | 73 | 60 | 4 | 2 | 186
  Transgender Spectrum | 1 | 5 | 0 | 0 | 0 | 6
  Not Reported | 1 | 1 | 0 | 0 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants] — Sex at birth.
  Participants
    Female | 4 | 12 | 11 | 2 | 1 | 30
    Male | 45 | 67 | 49 | 2 | 2 | 165
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 30 | 18 | 1 | 2 | 68
  Not Hispanic or Latino | 32 | 48 | 42 | 3 | 1 | 126
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 12 | 1 | 1 | 0 | 0 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 35 | 39 | 3 | 1 | 97
  White | 14 | 36 | 16 | 0 | 0 | 66
  More than one race | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 4 | 7 | 4 | 0 | 2 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 65 | 42 | 1 | 0 | 133
  Malawi | 4 | 3 | 3 | 0 | 1 | 11
  Brazil | 6 | 10 | 8 | 1 | 0 | 25
  Zimbabwe | 0 | 0 | 6 | 2 | 0 | 8
  Thailand | 12 | 1 | 0 | 0 | 0 | 13
  Peru | 2 | 0 | 1 | 0 | 2 | 5
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 22.5 [20.3 to 25.6] | 25.9 [21.4 to 28.8] | 23.8 [21.4 to 28.2] | 22.7 [17.7 to 28.4] | 23.2 [19.4 to 26.1] | 24.0 [21.2 to 28.0]
HIV-1 RNA (log10 copies per mL) [Median (Inter-Quartile Range); unit: log10(copies per mL)] — RNA levels below the lower limit of quantification (40 copies per mL) were imputed as 39 copies per mL.
  log10(copies per mL) | 6.4 [5.3 to 7.0] | 6.5 [6.0 to 7.0] | 5.4 [5.0 to 6.4] | 5.0 [3.0 to 6.3] | 1.6 [1.6 to 1.6] | 6.2 [5.2 to 6.8]
HIV-1 RNA [Count of Participants; unit: Participants]
  <40 copies per mL | 0 | 0 | 1 | 1 | 3 | 5
  40 - <1000 copies per mL | 1 | 0 | 0 | 0 | 0 | 1
  1000 - <10,000 copies per mL | 0 | 2 | 6 | 0 | 0 | 8
  10,000 - <100,000 copies per mL | 9 | 4 | 10 | 1 | 0 | 24
  100,000 - <1,000,000 copies per mL | 9 | 13 | 23 | 1 | 0 | 46
  1,000,000 - <10,000,000 copies per mL | 17 | 39 | 16 | 0 | 0 | 72
  >= 10,000,000 copies per mL | 13 | 21 | 4 | 1 | 0 | 39
CD4 Count [Median (Inter-Quartile Range); unit: cells per mm^3] — Population: Baseline CD4 measurements were not obtained for three participants.
  cells per mm^3
    number analyzed (Participants) | 48 | 78 | 60 | 4 | 2 | 192
    (all) | 348 [211 to 493] | 383 [264 to 538] | 490 [366 to 652] | 436 [401 to 647] | 1090 [604 to 1576] | 406 [284 to 575]
CD8 Count [Median (Inter-Quartile Range); unit: cells per mm^3] — Population: Baseline CD8 measurements were not obtained for seven participants.
  cells per mm^3
    number analyzed (Participants) | 47 | 76 | 59 | 4 | 2 | 188
    (all) | 322 [176 to 463] | 544 [309 to 923] | 1016 [766 to 1777] | 1401 [932 to 1843] | 474 [372 to 575] | 613 [336 to 1030]
Cell-associated HIV-1 DNA [Median (Inter-Quartile Range); unit: copies per 5 million CD4+ T-cells]
  Integrase Assay | 7739 [219 to 28351] | 15440 [3716 to 34658] | 10104 [1333 to 29716] | 4575 [0 to 9533] | 0 [0 to 0] | 10507 [1759 to 29499]
  Gag Assay | 4455 [1183 to 11782] | 6357 [2794 to 17213] | 5388 [2270 to 12938] | 3990 [1998 to 11000] | 0 [0 to 7] | 5586 [2219 to 13699]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Undetectable Cell-associated HIV-1 DNA (CAHD)
Description: Proportion of participants with 0 copies of CAHD per 5 million CD4+ blood-derived CD4+ T-cells (assayed by quantitative polymerase chain reaction [qPCR]), assessed separately and jointly by integrase and gag assays. In order for a participant to be considered as having 0 copies of CAHD for joint assays, the participant must be found to have an undetectable CAHD result from both integrase and gag assays. If all participants in both arms had undetectable CAHD then the statistical test was not performed.
Time Frame: At week 48
Population: Participants who maintained HIV-1 RNA<50 copies/mL at week 48 with no ART interruption of 7 or more consecutive days, no prior virologic failure (defined as having two consecutive HIV-1 RNA >200 copies/mL at week 24 or later or at any time after achieving HIV-1 RNA <50 copies/mL ), had available CAHD results from week 48 or week 49, and were enrolled during Fiebig Stage I-V.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm 1: Fiebig I/II | Arm 2: Fiebig III/IV | Arm 3: Fiebig V
Number analyzed (Participants) | 40 | 64 | 50
Proportion of participants
  Joint Assay (Integrase + Gag) | 0.00 [0.00 to 0.09] | 0.00 [0.00 to 0.06] | 0.00 [0.00 to 0.07]
  Integrase Assay | 0.10 [0.03 to 0.24] | 0.06 [0.02 to 0.15] | 0.10 [0.03 to 0.22]
  Gag Assay | 0.03 [0.00 to 0.13] | 0.02 [0.00 to 0.08] | 0.00 [0.00 to 0.07]
Statistical Analysis 1: Comparison: Arm 1: Fiebig I/II vs Arm 2: Fiebig III/IV; Results from Integrase Assay. Null Hypothesis: There is no difference between Arm 1 and Arm 2 in the proportion of participants with undetectable CA-DNA; Test type: Superiority; p = 0.48, Fisher Exact — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 2: Comparison: Arm 1: Fiebig I/II vs Arm 3: Fiebig V; Results from Integrase Assay. Null Hypothesis: There is no difference between Arm 1 and Arm 3 in the proportion of participants with undetectable CA-DNA; Test type: Superiority; p = 1, Fisher Exact — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 3: Comparison: Arm 2: Fiebig III/IV vs Arm 3: Fiebig V; Results from Integrase Assay. Null Hypothesis: There is no difference between Arm 2 and Arm 3 in the proportion of participants with undetectable CA-DNA; Test type: Superiority; p = 0.50, Fisher Exact — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 4: Comparison: Arm 1: Fiebig I/II vs Arm 2: Fiebig III/IV; Results from Gag Assay. Null Hypothesis: There is no difference between Arm 1 and Arm 2 in the proportion of participants with undetectable CA-DNA; Test type: Superiority; p = 1, Fisher Exact — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 5: Comparison: Arm 1: Fiebig I/II vs Arm 3: Fiebig V; Results from Gag Assay. Null Hypothesis: There is no difference between Arm 1 and Arm 3 in the proportion of participants with undetectable CA-DNA; Test type: Superiority; p = 0.44, Fisher Exact — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 6: Comparison: Arm 2: Fiebig III/IV vs Arm 3: Fiebig V; Results from Gag Assay. Null Hypothesis: There is no difference between Arm 2 and Arm 3 in the proportion of participants with undetectable CA-DNA; Test type: Superiority; p = 1, Fisher Exact — No adjustments for multiple comparisons. P-value based on two-sided test

2. Secondary Outcome: HIV-1-specific CD4+ and T-cell Responses to Nef, Gag, Pol and Env by Flow Cytometry
Description: Percent of HIV-1-specific CD4+ T-cells expressing any cytokine/marker (CD40L, CD107a, IFNg, MIP1B, TNFa) to each of the 4 protein stimulants (nef, gag, pol and env) by flow cytometry while HIV-1 RNA is suppressed on ART. The results for a specific participant are calculated by subtracting the corresponding background control value (media control). If the result would be less than zero after background subtraction, the result was set to zero.
  Cytokine/Marker Names: CD40 ligand (CD40L); Cluster of Differentiation 107a (CD107a); Interferon gamma (IFNg); Macrophage Inflammatory Protein beta (MIP1B); Tumor Necrosis Factor alpha (TNFa)
Time Frame: At week 48
Population: Participants who maintained HIV-1 RNA<50 copies/mL at week 48 with no ART interruption of 7 or more consecutive days, no prior virologic failure (defined as having two consecutive HIV-1 RNA >200 copies/mL at week 24 or later or at any time after achieving HIV-1 RNA <50 copies/mL ), had available CAHD results from week 48 or week 49, had available immunology marker results where active control result is greater than or equal to the media control, and were enrolled during Fiebig Stage I-V.
Measure: Median (Inter-Quartile Range); unit: Percentage of CD4+ T-cells
Arm/Group | Arm 1: Fiebig I/II | Arm 2: Fiebig III/IV | Arm 3: Fiebig V
Number analyzed (Participants) | 37 | 60 | 46
Percentage of CD4+ T-cells
  CD4+ T-cell Response to Env | 0.00 [0.00 to 0.24] | 0.00 [0.00 to 0.09] | 0.08 [0.00 to 0.17]
  CD4+ T-cell Response to Gag | 0.06 [0.00 to 0.23] | 0.19 [0.03 to 0.31] | 0.14 [0.05 to 0.27]
  CD4+ T-cell Response to Nef | 0.04 [0.00 to 0.15] | 0.10 [0.00 to 0.26] | 0.10 [0.00 to 0.23]
  CD4+ T-cell Response to Pol | 0.00 [0.00 to 0.03] | 0.04 [0.00 to 0.13] | 0.04 [0.00 to 0.19]
Statistical Analysis 1: Comparison: Arm 1: Fiebig I/II vs Arm 2: Fiebig III/IV; Null Hypothesis: There is no difference between Arm 1 and Arm 2 in percentage of HIV-1-specific CD4+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Env protein stimulant; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 2: Comparison: Arm 1: Fiebig I/II vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 1 and Arm 3 in percentage of HIV-1-specific CD4+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Env protein stimulant; Test type: Superiority; p = 0.46, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 3: Comparison: Arm 2: Fiebig III/IV vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 2 and Arm 3 in percentage of HIV-1-specific CD4+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Env protein stimulant; Test type: Superiority; p = 0.056, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 4: Comparison: Arm 1: Fiebig I/II vs Arm 2: Fiebig III/IV; Null Hypothesis: There is no difference between Arm 1 and Arm 2 in percentage of HIV-1-specific CD4+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Gag protein stimulant; Test type: Superiority; p = 0.025, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 5: Comparison: Arm 1: Fiebig I/II vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 1 and Arm 3 in percentage of HIV-1-specific CD4+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Gag protein stimulant; Test type: Superiority; p = 0.072, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 6: Comparison: Arm 2: Fiebig III/IV vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 2 and Arm 3 in percentage of HIV-1-specific CD4+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Gag protein stimulant; Test type: Superiority; p = 0.47, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 7: Comparison: Arm 1: Fiebig I/II vs Arm 2: Fiebig III/IV; Null Hypothesis: There is no difference between Arm 1 and Arm 2 in percentage of HIV-1-specific CD4+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Nef protein stimulant; Test type: Superiority; p = 0.086, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 8: Comparison: Arm 1: Fiebig I/II vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 1 and Arm 3 in percentage of HIV-1-specific CD4+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Nef protein stimulant; Test type: Superiority; p = 0.18, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 9: Comparison: Arm 2: Fiebig III/IV vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 2 and Arm 3 in percentage of HIV-1-specific CD4+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Nef protein stimulant; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 10: Comparison: Arm 1: Fiebig I/II vs Arm 2: Fiebig III/IV; Null Hypothesis: There is no difference between Arm 1 and Arm 2 in percentage of HIV-1-specific CD4+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Pol protein stimulant; Test type: Superiority; p = 0.061, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 11: Comparison: Arm 1: Fiebig I/II vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 1 and Arm 3 in percentage of HIV-1-specific CD4+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Pol protein stimulant; Test type: Superiority; p = 0.042, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 12: Comparison: Arm 2: Fiebig III/IV vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 2 and Arm 3 in percentage of HIV-1-specific CD4+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Pol protein stimulant; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test

3. Secondary Outcome: HIV-1-specific CD8+ and T-cell Responses to Nef, Gag, Pol and Env by Flow Cytometry
Description: Percent of HIV-1-specific CD8+ T-cells expressing any cytokine/marker (CD40L, CD107a, IFNg, MIP1B, TNFa) to each of the 4 protein stimulants (nef, gag, pol and env) by flow cytometry while HIV-1 RNA is suppressed on ART. The results for a specific participant are calculated by subtracting the corresponding background control value (media control). If the result would be less than zero after background subtraction, the result was set to zero.
  Cytokine/Marker Names: CD40 ligand (CD40L); Cluster of Differentiation 107a (CD107a); Interferon gamma (IFNg); Macrophage Inflammatory Protein beta (MIP1B); Tumor Necrosis Factor alpha (TNFa)
Time Frame: At 48 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percentage of CD8+ T-cells
Arm/Group | Arm 1: Fiebig I/II | Arm 2: Fiebig III/IV | Arm 3: Fiebig V
Number analyzed (Participants) | 37 | 60 | 46
Percentage of CD8+ T-cells
  CD8+ T-cell Response to Env | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.08] | 0.00 [0.00 to 0.36]
  CD8+ T-cell Response to Gag | 0.15 [0.00 to 0.36] | 0.33 [0.06 to 0.67] | 0.28 [0.00 to 0.61]
  CD8+ T-cell Response to Nef | 0.03 [0.00 to 0.32] | 0.15 [0.00 to 0.44] | 0.33 [0.04 to 0.68]
  CD8+ T-cell Response to Pol | 0.00 [0.00 to 0.08] | 0.05 [0.00 to 0.23] | 0.08 [0.00 to 0.26]
Statistical Analysis 1: Comparison: Arm 1: Fiebig I/II vs Arm 2: Fiebig III/IV; Null Hypothesis: There is no difference between Arm 1 and Arm 2 in percentage of HIV-1-specific CD8+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Env protein stimulant; Test type: Superiority; p = 0.97, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 2: Comparison: Arm 1: Fiebig I/II vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 1 and Arm 3 in percentage of HIV-1-specific CD8+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Env protein stimulant; Test type: Superiority; p = 0.21, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 3: Comparison: Arm 2: Fiebig III/IV vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 2 and Arm 3 in percentage of HIV-1-specific CD8+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Env protein stimulant; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 4: Comparison: Arm 1: Fiebig I/II vs Arm 2: Fiebig III/IV; Null Hypothesis: There is no difference between Arm 1 and Arm 2 in percentage of HIV-1-specific CD8+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Gag protein stimulant; Test type: Superiority; p = 0.055, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 5: Comparison: Arm 1: Fiebig I/II vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 1 and Arm 3 in percentage of HIV-1-specific CD8+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Gag protein stimulant; Test type: Superiority; p = 0.28, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 6: Comparison: Arm 2: Fiebig III/IV vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 2 and Arm 3 in percentage of HIV-1-specific CD8+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Gag protein stimulant; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 7: Comparison: Arm 1: Fiebig I/II vs Arm 2: Fiebig III/IV; Null Hypothesis: There is no difference between Arm 1 and Arm 2 in percentage of HIV-1-specific CD8+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Nef protein stimulant; Test type: Superiority; p = 0.35, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 8: Comparison: Arm 1: Fiebig I/II vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 1 and Arm 3 in percentage of HIV-1-specific CD8+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Nef protein stimulant; Test type: Superiority; p = 0.007, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 9: Comparison: Arm 2: Fiebig III/IV vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 2 and Arm 3 in percentage of HIV-1-specific CD8+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Nef protein stimulant; Test type: Superiority; p = 0.045, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 10: Comparison: Arm 1: Fiebig I/II vs Arm 2: Fiebig III/IV; Null Hypothesis: There is no difference between Arm 1 and Arm 2 in percentage of HIV-1-specific CD8+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Pol protein stimulant; Test type: Superiority; p = 0.085, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 11: Comparison: Arm 1: Fiebig I/II vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 1 and Arm 3 in percentage of HIV-1-specific CD8+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Pol protein stimulant; Test type: Superiority; p = 0.044, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 12: Comparison: Arm 2: Fiebig III/IV vs Arm 3: Fiebig V; Null Hypothesis: There is no difference between Arm 2 and Arm 3 in percentage of HIV-1-specific CD8+ T-cells expressing any cytokine (CD40L, CD107a, IFNg, MIP1B, TNFa) in response to Pol protein stimulant; Test type: Superiority; p = 0.60, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons. P-value based on two-sided test

4. Secondary Outcome: Proportion of Participants With Undetectable Cell-associated HIV-1 DNA (CAHD) Prior to ART Initiation
Description: Proportion of participants with 0 copies of CAHD per million CD4+ blood-derived CD4+ T-cells (assayed by quantitative PCR [qPCR]), assessed separately and jointly by integrase and gag assays. In order for a participant to be considered as having 0 copies of CAHD for joint assays, the participant must be found to have an undetectable CAHD result from both integrase and gag assays. If all participants in both arms had undetectable CAHD then the statistical test was not performed.
Time Frame: At week 0
Population: All participants who enrolled during Fiebig Stage I-V and had available CAHD at week 0.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm 1: Fiebig I/II | Arm 2: Fiebig III/IV | Arm 3: Fiebig V
Number analyzed (Participants) | 48 | 78 | 60
Proportion of participants
  Joint Assay (Integrase + Gag) | 0.00 [0.00 to 0.07] | 0.01 [0.00 to 0.07] | 0.00 [0.00 to 0.06]
  Integrase Assay | 0.04 [0.01 to 0.14] | 0.03 [0.00 to 0.09] | 0.07 [0.02 to 0.16]
  Gag Assay | 0.00 [0.00 to 0.07] | 0.01 [0.00 to 0.07] | 0.00 [0.00 to 0.06]
Statistical Analysis 1: Comparison: Arm 1: Fiebig I/II vs Arm 2: Fiebig III/IV; Results from Joint Assay. Null Hypothesis: There is no difference between Arm 1 and Arm 2 in the proportion of participants with undetectable CA-DNA; Test type: Superiority; p = 1, Fisher Exact — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 2: Comparison: Arm 2: Fiebig III/IV vs Arm 3: Fiebig V; Results from Joint Assay. Null Hypothesis: There is no difference between Arm 2 and Arm 3 in the proportion of participants with undetectable CA-DNA; Test type: Superiority; p = 1, Fisher Exact — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 3: Comparison: Arm 1: Fiebig I/II vs Arm 2: Fiebig III/IV; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.64, Fisher Exact — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 4: Comparison: Arm 1: Fiebig I/II vs Arm 3: Fiebig V; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.69, Fisher Exact — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 5: Comparison: Arm 2: Fiebig III/IV vs Arm 3: Fiebig V; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.40, Fisher Exact — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 6: Comparison: Arm 1: Fiebig I/II vs Arm 2: Fiebig III/IV; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 1, Fisher Exact — No adjustments for multiple comparisons. P-value based on two-sided test
Statistical Analysis 7: Comparison: Arm 2: Fiebig III/IV vs Arm 3: Fiebig V; [analysis description as in outcome 1, analysis 6]; Test type: Superiority; p = 1, Fisher Exact — No adjustments for multiple comparisons. P-value based on two-sided test

ADVERSE EVENTS:
Time Frame: Step 1: From study entry to Step 1 Week 72, Step 2 entry, or premature study discontinuation on Step 1. Step 2: From step 2 entry to Step 2 Week 144 or premature study discontinuation on Step 2.
Description: All Grade ≥3 signs and symptoms, Grade ≥2 laboratory findings, all targeted diagnoses, adverse events (AEs) that led to a change in study treatment/intervention regardless of grade, and all AEs meeting serious adverse event (SAE) definition or expediated adverse event (EAE) reporting requirement were collected. The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, corrected Version 2.1, July 2017 was used. Fiebig VI/HIV Negative could not enroll to Step 2.
Groups:
- Step 1 Arm 1: Fiebig I/II: Participants enrolled during Fiebig stages I or II (non-reactive HIV-1 antibody).
  elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide or bictegravir/emtricitabine/tenofovir alafenamide or other medically-appropriate FDA-approved antiretroviral therapy: Participants received one tablet of elvitegravir 150mg/cobicistat 150mg/emtricitabine 200mg/tenofovir alafenamide 10mg by mouth daily with food or one tablet of bictegravir 50mg/emtricitabine 200mg/tenofovir alafenamide 25mg by mouth daily with or without food. Other non-study-provided ARV regimens were allowed for participants who were pregnant, breastfeeding, or unable/unwilling to take EVG/COBI/FTC/TAF or BIC/FTC/TAF, or for participants whose local health care/primary care provider preferred starting a different initial ARV regimen.
- Step 1 Arm 2: Fiebig III/IV: Participants enrolled during Fiebig stages III or IV (reactive HIV-1 antibody and negative or indeterminate results on the Western blot or Geenius HIV-1/HIV-2).
  elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide or bictegravir/emtricitabine/tenofovir alafenamide or other medically-appropriate FDA-approved antiretroviral therapy: Participants received one tablet of elvitegravir 150mg/cobicistat 150mg/emtricitabine 200mg/tenofovir alafenamide 10mg by mouth daily with food or one tablet of bictegravir 50mg/emtricitabine 200mg/tenofovir alafenamide 25mg by mouth daily with or without food. Other non-study-provided ARV regimens were allowed for participants who were pregnant, breastfeeding, or unable/unwilling to take EVG/COBI/FTC/TAF or BIC/FTC/TAF, or for participants whose local health care/primary care provider preferred starting a different initial ARV regimen.
- Step 1 Arm 3: Fiebig V: Participants enrolled during Fiebig stage V (reactive HIV-1 antibody and positive Western blot or Geenius HIV-1/HIV-2 without p31 band).
  elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide or bictegravir/emtricitabine/tenofovir alafenamide or other medically-appropriate FDA-approved antiretroviral therapy: Participants received one tablet of elvitegravir 150mg/cobicistat 150mg/emtricitabine 200mg/tenofovir alafenamide 10mg by mouth daily with food or one tablet of bictegravir 50mg/emtricitabine 200mg/tenofovir alafenamide 25mg by mouth daily with or without food. Other non-study-provided ARV regimens were allowed for participants who were pregnant, breastfeeding, or unable/unwilling to take EVG/COBI/FTC/TAF or BIC/FTC/TAF, or for participants whose local health care/primary care provider preferred starting a different initial ARV regimen.
- Step 1 Fiebig VI: Participants enrolled during Fiebig stage VI (reactive HIV-1 antibody and positive Western blot or Geenius HIV-1/HIV-2 without p31 band).
  elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide or bictegravir/emtricitabine/tenofovir alafenamide or other medically-appropriate FDA-approved antiretroviral therapy: Participants received one tablet of elvitegravir 150mg/cobicistat 150mg/emtricitabine 200mg/tenofovir alafenamide 10mg by mouth daily with food or one tablet of bictegravir 50mg/emtricitabine 200mg/tenofovir alafenamide 25mg by mouth daily with or without food. Other non-study-provided ARV regimens were allowed for participants who were pregnant, breastfeeding, or unable/unwilling to take EVG/COBI/FTC/TAF or BIC/FTC/TAF, or for participants whose local health care/primary care provider preferred starting a different initial ARV regimen.
- Step1 HIV Negative: Participants found to be HIV negative following the results of HIV-1 RNA testing at study entry. No study treatment.
- Step 2 Arm 1: Fiebig I/II: Participants enrolled during Fiebig stages I or II (non-reactive HIV-1 antibody) that enrolled to Step 2.
  elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide or bictegravir/emtricitabine/tenofovir alafenamide or other medically-appropriate FDA-approved antiretroviral therapy: Participants received one tablet of elvitegravir 150mg/cobicistat 150mg/emtricitabine 200mg/tenofovir alafenamide 10mg by mouth daily with food or one tablet of bictegravir 50mg/emtricitabine 200mg/tenofovir alafenamide 25mg by mouth daily with or without food. Other non-study-provided ARV regimens were allowed for participants who were pregnant, breastfeeding, or unable/unwilling to take EVG/COBI/FTC/TAF or BIC/FTC/TAF, or for participants whose local health care/primary care provider preferred starting a different initial ARV regimen.
- Step 2 Arm 2: Fiebig III/IV: Participants enrolled during Fiebig stages III or IV (reactive HIV-1 antibody and negative or indeterminate results on the Western blot or Geenius HIV-1/HIV-2) that enrolled to Step 2.
  elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide or bictegravir/emtricitabine/tenofovir alafenamide or other medically-appropriate FDA-approved antiretroviral therapy: Participants received one tablet of elvitegravir 150mg/cobicistat 150mg/emtricitabine 200mg/tenofovir alafenamide 10mg by mouth daily with food or one tablet of bictegravir 50mg/emtricitabine 200mg/tenofovir alafenamide 25mg by mouth daily with or without food. Other non-study-provided ARV regimens were allowed for participants who were pregnant, breastfeeding, or unable/unwilling to take EVG/COBI/FTC/TAF or BIC/FTC/TAF, or for participants whose local health care/primary care provider preferred starting a different initial ARV regimen.
- Step 2 Arm 3: Fiebig V: Participants enrolled during Fiebig stage V (reactive HIV-1 antibody and positive Western blot or Geenius HIV-1/HIV-2 without p31 band) that enrolled to Step 2.
  elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide or bictegravir/emtricitabine/tenofovir alafenamide or other medically-appropriate FDA-approved antiretroviral therapy: Participants received one tablet of elvitegravir 150mg/cobicistat 150mg/emtricitabine 200mg/tenofovir alafenamide 10mg by mouth daily with food or one tablet of bictegravir 50mg/emtricitabine 200mg/tenofovir alafenamide 25mg by mouth daily with or without food. Other non-study-provided ARV regimens were allowed for participants who were pregnant, breastfeeding, or unable/unwilling to take EVG/COBI/FTC/TAF or BIC/FTC/TAF, or for participants whose local health care/primary care provider preferred starting a different initial ARV regimen.
Arm/Group | Step 1 Arm 1: Fiebig I/II | Step 1 Arm 2: Fiebig III/IV | Step 1 Arm 3: Fiebig V | Step 1 Fiebig VI | Step1 HIV Negative | Step 2 Arm 1: Fiebig I/II | Step 2 Arm 2: Fiebig III/IV | Step 2 Arm 3: Fiebig V
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/79 | 0/60 | 0/4 | 0/3 | 1/26 | 0/42 | 0/23
Serious Adverse Events (participants affected / at risk) | 5/49 | 7/79 | 4/60 | 0/4 | 0/3 | 6/26 | 4/42 | 3/23
Other Adverse Events (participants affected / at risk) | 48/49 | 67/79 | 50/60 | 4/4 | 2/3 | 18/26 | 30/42 | 15/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 Arm 1: Fiebig I/II (N=49) | Step 1 Arm 2: Fiebig III/IV (N=79) | Step 1 Arm 3: Fiebig V (N=60) | Step 1 Fiebig VI (N=4) | Step1 HIV Negative (N=3) | Step 2 Arm 1: Fiebig I/II (N=26) | Step 2 Arm 2: Fiebig III/IV (N=42) | Step 2 Arm 3: Fiebig V (N=23)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fascial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Monkeypox (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Secondary syphilis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis B surface antigen positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cervical cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vascular skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Step 1 Arm 1: Fiebig I/II (N=49) | Step 1 Arm 2: Fiebig III/IV (N=79) | Step 1 Arm 3: Fiebig V (N=60) | Step 1 Fiebig VI (N=4) | Step1 HIV Negative (N=3) | Step 2 Arm 1: Fiebig I/II (N=26) | Step 2 Arm 2: Fiebig III/IV (N=42) | Step 2 Arm 3: Fiebig V (N=23)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thalassaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anogenital dysplasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute hepatitis C (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal chlamydia infection (Infections and infestations) | 4 | 0 | 2 | 0 | 0 | 5 | 2 | 0
Anal gonococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacterial diarrhoea (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Balanitis candida (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Chlamydial cervicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epididymitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Genital herpes simplex (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Genitourinary chlamydia infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Genitourinary tract gonococcal infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis A (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex anorectal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Latent syphilis (Infections and infestations) | 4 | 2 | 1 | 0 | 0 | 4 | 4 | 0
Latent tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Monkeypox (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neurosyphilis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal gonococcal infection (Infections and infestations) | 4 | 1 | 3 | 0 | 0 | 1 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngeal chlamydia infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Primary syphilis (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 2 | 2 | 0
Proctitis chlamydial (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 1 | 4 | 4
Proctitis gonococcal (Infections and infestations) | 1 | 3 | 3 | 0 | 0 | 1 | 0 | 0
Scabies (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Secondary syphilis (Infections and infestations) | 4 | 5 | 3 | 0 | 0 | 2 | 2 | 0
Shigella infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syphilis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syphilis genital (Infections and infestations) | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tonsillitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Trichomoniasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tubo-ovarian abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Urethritis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urethritis chlamydial (Infections and infestations) | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0
Urethritis gonococcal (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urethritis ureaplasmal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginitis gonococcal (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 5 | 2 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 5 | 4 | 0 | 0 | 0 | 0 | 1
Bilirubin conjugated increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0
Blood creatine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 16 | 23 | 16 | 0 | 0 | 2 | 4 | 4
Blood glucose decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 3 | 1 | 0 | 0 | 0 | 2 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chlamydia test positive (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 37 | 61 | 45 | 4 | 2 | 0 | 9 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 5 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Neisseria test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syphilis test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Trichomonal test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tuberculin test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitated depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Penile discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Essential hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 2 | 1 | 1 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (3):
  • Study Protocol (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT02859558/Prot_001.pdf
  • Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT02859558/SAP_002.pdf
  • Informed Consent Form (2016-06-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT02859558/ICF_000.pdf